CLINICAL TRIAL: NCT00221130
Title: Clinical Trial of Regenerative Periodontal Tissue by Transplanting Mesenchymal Stem Cells and Osteoblast Cells - I, II Phase-
Brief Title: Clinical Trials of Regeneration for Periodontal Tissue
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: ArBlast Co.,Ltd. (Industry); Nagoya University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRI PDT03-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Adult Periodontitis
Keywords: Regenerative medicine; Periodontal tissue
MeSH Terms: conditions — Chronic Periodontitis

INTERVENTIONS:
Procedure: surgical operation of cell transplantation

SUMMARY:
Adult periodontitis is a chronic infective disease affecting the periodontium. Periodontitis induce the destruction of attachment apparatus of teeth, resulting in periodontal pocket formation and teeth loss. This study will test the safety and efficacy of alveolous bone reproduction by the transplantation of mixture named periodontium injectable gel for the adult periodontitis patients. Injectable gel is the mixture of ex-vivo cultured mesenchymal stem stem cells, ex-vivo cultured osteoblast-like cells differentiated from mesenchymal stem cells and scaffold (include, platelet rich plasma, human thrombin and calcium chloride).

DETAILED DESCRIPTION:
Periodontal disease is an infectious disease. Gingivitis and periodontitis are the 2 major forms of this. Their primary etiology is bacterial plaque, which can induce destruction of the periodontal apparatus. Gingivitis is inflammation of the gingival that does not result in clinical attachment loss. Periodontitis is inflammation of the gingival and is characterized by loss of connective tissue attachment and alveolar bone.

Therapeutic approaches for periodontitis are divided into two categories: 1) anti-infective treatment; 2) regenerative therapy.

Several surgical techniques have been developed to regenerate periodontal tissues including guided tissue regeneration, bone grafting, the use of enamel matrix derivative. However, these techniques are not reached for complete regeneration of the periodontium.

This study will test the safety and efficacy of alveolous bone reproduction by the transplantation of mixture named periodontium injectable gel for the adult periodontitis patients. Injectable gel is the mixture of ex-vivo cultured mesenchymal stem stem cells, ex-vivo cultured osteoblast-like cells differentiated from mesenchymal stem cells and scaffold (include, platelet rich plasma, human thrombin and calcium chloride).

ELIGIBILITY:
Inclusion Criteria:

* 1.Patient with adult periodontitis. 2. There are ４mm or more pocket using . 3.There are ten existing tooth or more of the lower jaw. 4.The brushing instruction is received, and the plaque control is maintained excellently. 5.The recovery by an existing periodontal operation cannot be expected. 6.The age is from 35 to 60 years old. 7.Blood clot function is normal. 8.The liver function is normal. 9.The intention and the ability of going to hospital regularly are possessed. 10.Agreement by the document is obtained.

Exclusion Criteria:

* 1.Patient who has acute symptom of periodontitis. 2.Patient that decayed tooth is on teeth or the next teeth to be treated. 3.Patient who has contracted diabetic or autoimmune disease. 4.Patient who has contracted infectious disease. 5.Patient who has contracted osteoporosis. 6.Patient who has smoking habit within six months before it registers. 7.Patient who is taking treatment of hypertension and/or epilepsy. 8.Patient who has pregnancy or doubt of pregnancy. 9.Patient who has heavy allergic disease.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2004-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Alveolar bone defect

SECONDARY OUTCOMES:
Tooth mobility

CONTACTS AND LOCATIONS:
Overall Officials: Shunsuke Baba, D.D.S, PhD, Principal Investigator — Ｉｎstitute of Biomedical Research and Innovation
Locations (1):
- Ｉｎstitute of Biomedical Research and Innovation, Kobe, Hyogo Pref., Japan